CLINICAL TRIAL: NCT06802887
Title: Long-term Treatment With Ustekinumab in Patients With Crohn's Disease and Ulcerative Colitis: a Monocentric, Observational, Retrospective/Prospective Cohort Study
Brief Title: Long-term Treatment With Ustekinumab in Patients With Crohn's Disease and Ulcerative Colitis: a Cohort Study
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: USK-IBD
Record Dates: First submitted 2024-12-01; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-10

CONDITIONS: IBD - Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Monocentric observational retrospective/prospective pharmacological study. Clinical records of patients with Ulcerative Colitis and Crohn's Disease who started therapy with Ustekinumab between February 2019 and March 2021 at the IBD Unit will be reviewed. The main objective is to evaluate the overall persistence of patients with Crohn's Disease and Ulcerative Colitis who started Ustekinumab between February 2019 and March 2021, as well as the impact of treatment on the natural history of the disease. The study involves the collection of follow-up data for a maximum period of 24 months from the start of therapy. For patients who began therapy with Ustekinumab from February 2019 up to 24 months before the start of enrollment, data collection will be conducted retrospectively. For patients who have undergone therapy with Ustekinumab within 24 months prior to the start of enrollment, and up to March 2021, data will be collected both retrospectively and prospectively.

DETAILED DESCRIPTION:
The medical records of patients with Crohn's Disease and Ulcerative Colitis who started therapy with Ustekinumab between February 2019 and March 2021 have been selected. Initially, it was estimated that approximately 350 patients would be eligible for enrollment in the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Male and female patients, aged ≥18 years
* Patients who began treatment with Ustekinumab according to the indications for marketing authorization, following clinical practice and the information contained in the product's technical data sheet, during the period from February 2019 to March 2021.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is expected to enroll approximately 300 patients with Crohn's Disease and 50 patients with Ulcerative Colitis who started therapy with Ustekinumab during the period from February 2019 to March 2021, as part of the normal care pathway, at the Regional Reference Center for Inflammatory Bowel Diseases in Emilia-Romagna.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2021-07-18 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Overall persistence of patients with Crohn's Disease and Ulcerative Colitis who started Ustekinumab. | Baseline; through study completion, an average of 2 years
  Evaluate the percentage of treatment discontinuation; Evaluate the percentage of patients for whom therapy optimization was necessary through the reduction of the interval between administrations; Evaluate the percentage of patients for whom it was necessary to switch to another therapy;

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Gionchetti, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy